CLINICAL TRIAL: NCT01379768
Title: Polymorphonuclear Leukocyte Response During Overnight Lens Wear
Brief Title: Study of the Cell Response in the Tear Film After Overnight Contact Lens Wear
Acronym: CORNWALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P-373-C-102
Record Dates: First submitted 2011-06-09; First posted 2011-06-23 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: White Blood Cells

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lotrafilcon A (Active Comparator): Lotrafilcon A contact lenses worn on a daily wear basis for 1 week, followed by 8 hours overnight wear in a replacement pair. After a 12-hour washout period, a new pair of lotrafilcon A contact lenses were dispensed for 4 weeks of daily wear, followed by 8 hours overnight wear.
  Interventions: Device: Lotrafilcon A contact lens; Device: Clear Care Cleaning and Disinfection Solution
- Lotrafilcon B (Active Comparator): Lotrafilcon B contact lenses worn on a daily wear basis for 1 week, followed by 8 hours overnight wear in a replacement pair. After a 12-hour washout period, a new pair of lotrafilcon B contact lenses were dispensed for 4 weeks of daily wear, followed by 8 hours overnight wear.
  Interventions: Device: Lotrafilcon B contact lens; Device: Clear Care Cleaning and Disinfection Solution
- No lens wear (No Intervention): No contact lens wear for the duration of the study. One 8-hour sleep at 1 week, followed by an 8-hour sleep 4 weeks later.

INTERVENTIONS:
Device: Lotrafilcon A contact lens — Commercially marketed, silicone hydrogel, single-vision contact lens FDA-approved for daily and extended (overnight) wear for up to 30 nights.
  Other Names: AIR OPTIX NIGHT & DAY AQUA
  Arms: Lotrafilcon A
Device: Lotrafilcon B contact lens — Commercially marketed, silicone hydrogel, single-vision contact lens FDA-approved for daily or extended (overnight) wear up to 6 nights.
  Other Names: NIGHT & DAY®
  Arms: Lotrafilcon B
Device: Clear Care Cleaning and Disinfection Solution — Hydrogen peroxide-based contact lens care system for nightly cleaning and disinfection of study lenses
  Other Names: Clear Care®
  Arms: Lotrafilcon A; Lotrafilcon B

SUMMARY:
The purpose of this study was to count and analyze the white blood cells in tear samples collected from study participants following sleep. The results from contact lens wearers were compared with the results from non-contact lens wearers.

DETAILED DESCRIPTION:
The objective of the study was to determine and compare the relative oxidative response of polymorphonuclear neutrophils (PMNs), the relative cell adhesion response of PMNs, and the leukocyte population in tear samples collected from contact lens wearers and non-contact lens wearers. Tear samples were collected via a binocular eye-wash. The samples were processed, and a cell count was performed using a hemacytometer. Flow cytometry was used to determine the expression of different PMN cell markers before and after stimulation with bacterial lipopolysaccharide (LPS).

ELIGIBILITY:
Inclusion Criteria:

* 17 years of age or older.
* Ocular examination in the last two years.
* Has up-to-date spectacles.
* Falls into one of the following three categories:

  * Adapted wearer of Lotrafilcon A contact lenses
  * Adapted wearer of Lotrafilcon B contact lenses
  * Does not wear contact lenses
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Ocular disease
* Systemic or topical medications that may affect ocular health.
* Known sensitivity to diagnostic pharmaceuticals used in study.
* Uses artificial tears and/or rewetting drops.
* Wears contact lenses on an overnight basis for more than one night per week.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom FAAO, Director, Principal Investigator — Centre for Contact Lens Research, School of Optometry, University of Waterloo
Locations (1):
- University of Waterloo Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from one study center located in Canada.
Period: Overall Study
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Started | 23 | 22 | 20
Completed | 20 | 21 | 20
Not Completed | 3 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear | Total
Number analyzed (Participants) | 23 | 22 | 20 | 65
Age, Customized [Median (Full Range); unit: years] | 22 [19 to 50] | 23.5 [19 to 50] | 23.5 [20 to 41] | 23 [19 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 13 | 49
  Male | 6 | 3 | 7 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 23 | 22 | 20 | 65

OUTCOME MEASURES:

1. Primary Outcome: Leukocyte Population
Description: A tear sample was collected after 8 hours of sleep using an ocular surface cell collection apparatus (OSCCA). Different types of white blood cells (leukocytes) were identified, which included neutrophils, monocytes, and lymphocytes. The total amount of leukocytes for contact lens wearers and non-lens wearers is presented. Potential differences in leukocyte count between lens wearers and non-lens wearers may indicate a different immune response.
Time Frame: Week 5
Population: This reporting group includes all participants who completed the study per protocol.
Measure: Mean (Standard Deviation); unit: Leukocytes
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Number analyzed (Participants) | 20 | 19 | 20
Leukocytes | 583187 (832636) | 420345 (355940) | 738140 (609853)

2. Primary Outcome: Relative Cell Adhesion Response of Polymorphonuclear Leukocytes (PMNs)
Description: A tear sample was collected after 8 hours of sleep using an ocular surface cell collection apparatus (OSCCA) and analyzed on a flow cytometer. CD54 is a protein typically found in the cell membrane of leukocytes, which up-regulates during inflammation and promotes cell adhesion. Cell adhesion response is reported as a ratio of stimulated to non-stimulated samples.
Time Frame: Week 5
Population: This reporting group includes all participants who completed the study per protocol.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Number analyzed (Participants) | 20 | 18 | 19
Ratio | 1.1 (0.2) | 1.2 (0.2) | 1.1 (0.1)

3. Primary Outcome: Relative Oxidative Response of Polymorphonuclear Leukocytes (PMNs)
Description: A tear sample was collected after 8 hours of sleep using an ocular surface cell collection apparatus (OSCCA) and analyzed on a flow cytometer. Oxidative response is reported as a ratio of activated to non-activated samples. DCF (dichlorofluorescein diacetate) is a molecular probe that measures the oxidative burst. Upon stimulation, the PMNs synthesize reactive oxygen species, such as superoxide or hydrogen peroxide, which is detected by the probe. Differences in the oxidative response between contact lens wearers and non-lens wearers is indicated by a shift in the ratio (stimulated/unstimulated).
Time Frame: Week 5
Population: This reporting group includes all participants who completed the study per protocol.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Number analyzed (Participants) | 20 | 19 | 20
Ratio | 1.2 (0.5) | 1.7 (1.1) | 1.3 (0.6)

4. Primary Outcome: Change From Week 1 in Leukocyte Population at Week 5
Description: A tear sample was collected after 8 hours of sleep using an ocular surface cell collection apparatus (OSCCA). Different types of white blood cells (leukocytes) were identified, which included neutrophils, monocytes, and lymphocytes. The difference between total leukocytes for contact lens wearers and non-lens wearers (Week 5 minus Week 1) is presented.
Time Frame: Week 1, Week 5
Population: This reporting group includes all participants who completed the study per protocol.
Measure: Mean (Standard Deviation); unit: Leukocytes
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Number analyzed (Participants) | 19 | 19 | 19
Leukocytes | -1377 (453,119) | -95301 (632752) | 122316 (519976)

5. Primary Outcome: Change From 1 Week in Relative Cell Adhesion Response of PMNs at Week 5
Description: A tear sample was collected after 8 hours of sleep using an ocular surface cell collection apparatus (OSCCA) and analyzed on a flow cytometer. Cell adhesion response is reported as a ratio of activated to non-activated samples. The difference between the ratio data for contact lens wearers and non-lens wearers (Week 5 minus Week 1) is presented.
Time Frame: Week 1, Week 5
Population: This reporting group includes all participants who completed the study per protocol.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Number analyzed (Participants) | 18 | 15 | 16
Ratio | -0.01 (0.23) | 0.00 (0.24) | -0.01 (0.20)

6. Primary Outcome: Change From Week 1 in Relative Oxidative Response of PMNs at Week 5
Description: A tear sample was collected after 8 hours of sleep using an ocular surface cell collection apparatus (OSCCA) and analyzed on a flow cytometer. Oxidative response is reported as a ratio of activated to non-activated samples. The difference between the ratio data for contact lens wearers and non-lens wearers (Week 5 minus Week 1) is presented.
Time Frame: Week 1, Week 5
Population: This reporting group includes all participants who completed the study per protocol.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Number analyzed (Participants) | 19 | 18 | 19
Ratio | 0.05 (0.94) | 0.24 (1.20) | -0.19 (0.58)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study.
Description: This reporting group includes all enrolled participants.
Arm/Group | Lotrafilcon A | Lotrafilcon B | No Lens Wear
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.